CLINICAL TRIAL: NCT03469076
Title: Studie Van de Huidmicrobiota en Het Potentieel Van Een crème Met Probiotica Bij Personen Met Acne
Brief Title: Studying the Skin Microbiome and the Potential of a Topical Probiotic Cream for Patients With Acne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité, UZA, Prof. Julien Lambert, MD, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16/14/168; B300201628507 (Other: Belgian Registration)
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Acne Vulgaris
Keywords: Acne, Comedonal, Mild to Moderate Papulopustular Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACN Cream (Experimental): Patients with mild to moderate acne using ACN Cream
  Interventions: Other: YUN ACN Cream

INTERVENTIONS:
Other: YUN ACN Cream — YUN ACN Cream with live probiotic bacteria (min. 10-6 à 10-7 CFU per application) applied twice daily (morning and evening) on the entire face
  Other Names: topical cream with live probiotic bacteria

SUMMARY:
In this study the topical use of cream with live probiotic bacteria was evaluated for its efficacy in reducing acne symptoms and its effect on the skin microbiota on patients with acne. Patients with mild to moderate acne used the probiotic cream for 8 weeks and clinical evaluation and sampling was done at start, 4, 8 and 10 weeks. Next-Generation Sequencing was used to analyze the skin microbiota of the patients.

DETAILED DESCRIPTION:
Probiotics are live micro-organisms which when administered in adequate amounts can exert a health benefit on the host. This health-promoting effects have been extensively studied in the gastrointestinal niche but it becomes more and more clear that other niches are also interesting for the potential of probiotics. Recent breakthroughs in 'next generation sequencing' (NGS) technologies are making it now possible to map the microbiota after DNA extraction, which is very interesting for bacteria that are not or difficult to cultivate. The research into the microbiota of the skin with such new NGS technologies currently limited, but shows that there is also an equilibrium in the skin composition of the microbiota and that there is a disturbance of the skin microbiota in acne (Murillo & Raoult, 2013). In acne vulgaris it is known that the condition is multifactorial and that both hormonal triggers and environmental factors play a role. However, it is also known that Propionibacterium acnes play an important role in the inflammation of the sebaceous gland follicles. Probiotic strains with antipathogenic activity against this bacterium and suitable for application to the skin is thus potentially able to restore the balance of the skin microbiota and reduce acne symptoms.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate acne

Exclusion Criteria:

* local treatments, including cleansers, soaps, antimycotics and antibiotics within 2 weeks prior to start of study
* use of oral antibiotics within 4 weeks prior to start of study
* use of systemic retinoids within 6 months prior to start of study

Ages: 12 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04-25 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Skin microbiome differences | baseline; after 4 and 8 weeks of treatment; at 10 weeks, i.e. 2 weeks after stop of treatment
  Analysis of the skin's microbiome at start (baseline) and after treatment with the ACN Cream
Clinical acne symptoms | baseline, at 4, 8 and 10 weeks
  Clinical evaluation of acne symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Julien Lambert, Prof. dr, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital, Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided